CLINICAL TRIAL: NCT00718731
Title: Ascending Single Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GSI 136 Administered Orally to Healthy Young and Healthy Elderly Subjects
Brief Title: Study GSI-136 in Healthy Young and Healthy Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Wyeth
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3225A1-1000
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-04

CONDITIONS: Alzheimer Disease; Healthy
Keywords: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Subject on active drug
  Interventions: Drug: GSI-136
- 2 (Placebo Comparator): Subject on placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GSI-136
  Arms: 1
Other: Placebo
  Arms: 2

SUMMARY:
This is a first-in-humans study of GSI-136, a drug being developed for the treatment of Alzheimer Disease. The main purpose of this study is to determine whether GSI-136 is safe and tolerable in healthy young and healthy elderly subjects. The amount of drug in the body and the effects of the drug on the body will also be evaluated at certain timepoints.

ELIGIBILITY:
<Inclusion:

1. Men or women of nonchildbearing potential (WONCBP) aged 18 to 50 years or greater than 65 years, inclusive, at screening. WONCBP may be included if they are either surgically sterile (hysterectomy and/or oophorectomy) or postmenopausal for greater than 1 year (with follicle-stimulating hormone [FSH] level greater than 38 mIU/mL) and must have a negative pregnancy test result within 48 hours before test article administration. Women who are surgically sterile must provide documentation of the procedure by an operative report or by ultrasound scan. Sexually active men must agree to use a medically acceptable form of contraception during the study and continue it for 12 weeks after test article administration.
2. Body mass index (BMI) in the range of 18.0 to 30.0 kg/m2 and body weight greater than 50 kg.

3) The elderly subjects must be generally healthy, but may be enrolled with a stable, chronic illness, if it is well controlled and does not interfere with the primary objective of the study. Subjects may be included with clinically important deviations from normal limits in medical history, physical examination findings, vital sign measurements, 12-lead ECGs, or clinical laboratory test results that are associated with stable, chronic, and well-controlled medical conditions.

Exclusion:

1. Any history or presence of chronic respiratory disorder or disease including but not limited to asthma, sleep apnea, or chronic obstructive pulmonary disease (COPD).
2. Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
3. Presence or history of thyroid disease, symptomatic vertigo, significant cardiac valvular disease, congestive heart failure, angina pectoris, significant cardiac arrhythmia, or seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of GSI-136 as evaluated from reported adverse events, scheduled physical examinations, vital sign measurements, orthostatic vital sign measurements, cardiac rhythm monitoring, 12-lead ECGs, and clinical laboratory test results. | 6 months

SECONDARY OUTCOMES:
Pharmacokinetics as evaluated from the blood and urine concentrations of GSI-136; Pharmacodynamics as evaluated from the levels of select biomarkers in the blood and the administration of a visual analog scale to measure sedation effects. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- New York, New York, United States